CLINICAL TRIAL: NCT06761300
Title: Psychological Assessment in Patients Suffering from Chronic Pain Treated with Spinal Cord Stimulation
Brief Title: Psychological Assessment in Patients Treated with Spinal Cord Stimulation
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 2028
Record Dates: First submitted 2024-11-25; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Stimulation (SCS); Chronic Pain
Keywords: Spinal Cord Stimulation; chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with chronic pain: Patients suffering from chronic pain treated with Spinal Cord Stimulation
  Interventions: Other: Psychological assessment

INTERVENTIONS:
Other: Psychological assessment — Psychological assessment evaluation at different time points and its correlation with pain outcomes and satisfaction with the SCS intervention.

SUMMARY:
This is a prospective observational study to investigate the impact of spinal cord stimulation (SCS) procedure in chronic pain perception and management. Patients' psychological status at different time points and its correlation with pain outcomes and satisfaction with the SCS intervention will be also evaluated.

The primary aim is to study the associations between psychological variables and intervention outcomes (pain reduction, satisfaction, removal of SCS). Our hypothesis is that people with higher scores in anxiety and depression symptoms would report lower satisfaction with SCS procedure and higher levels of perceived pain after the implantation of the device

DETAILED DESCRIPTION:
More than 30% of people worldwide suffer from chronic pain (CP), defined as "an unpleasant sensory and emotional experience associated with actual or potential tissue damage, or described in terms of such damage".

Patients suffering from CP in charge of the Palliative Care and Pain Therapy Division at the European Institute of Oncology IRCCS (Milan, Italy) will be proposed to undergo SCS surgical implantation to mitigate pain symptoms.

The SCS surgical implantation is a two-step procedure; after the hospital admission, a temporary SCS device will be firstly implanted. In this way patients have the possibility to experiment the device impact on their CP conditions, to familiarize with the external device and adjust to its presence, and to eventually grow their motivation toward the implantation of the permanent device. Only after one month, if the patients are convinced of the intervention utility, the temporary device will be changed with a permanent one.

After the medical consultation, patients accepting the surgical procedure and meeting the inclusion criteria will be invited to participate to the study.

Patients signing the Informed Consent will receive a link to complete a set of questionnaires investigating psychological well-being, the impact of chronic pain in daily activities and the decision-making process to undergo to a surgical procedure. Participants who will not be able to complete the online form, will fill it on paper. Patients will complete different questionnaires at different time-points before and after the two-step SCS implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering from chronic pain (VAS>4) from at least 6 months
2. Patient eligible for SCS implantation
3. Age >18 years old
4. Willingness and ability to comply with scheduled visits and other trial procedures
5. Understanding and speaking Italian language
6. Written informed consent

Exclusion Criteria:

1. Psychiatric disorders or conditions that might impair the ability to give informed consent
2. Comorbidity that may impact on compliance to study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from CP in charge of the Palliative Care and Pain Therapy Division at the European Institute of Oncology IRCCS (Milan, Italy) will be proposed to undergo SCS surgical implantation to mitigate pain symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-09 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pain reduction | 8 months
  The correlation between each psychological variable and pain reduction will be evaluated using the scores of the following validated questionnaires: State-Trait Anxiety Inventory (STAI-Y), Beck Depression Inventory II (BDI-II), Pain Resilience Scale (PRS), Pain Catastrophizing Scale (PCS), and Brief Pain Inventory (BPI) questionnaire. Details on measurement: The correlation will be evaluated using Pearson's correlation coefficient.
Evaluation of removal of SCS | 8 months
  The correlation between each psychological variable, pain reduction and removal of SCS will be evaluated using the scores of the following validated questionnaires: State-Trait Anxiety Inventory (STAI-Y), Beck Depression Inventory II (BDI-II), Pain Resilience Scale (PRS), Brief Pain Inventory (BPI) and Pain Catastrophizing Scale (PCS). Details on measurement: The correlation will be evaluated using Student's t-test.
Evaluation of satisfaction. | 8 months
  Patients SCS satisfaction and the correlation between each psychological variable will be evaluated using the scores of the following validated questionnaires: State-Trait Anxiety Inventory (STAI-Y), Beck Depression Inventory II (BDI-II), Pain Resilience Scale (PRS), Pain Catastrophizing Scale (PCS). Patients' satisfaction with the SCS procedure will be measured with the Patients Global Impression of Change (PGIC) questionnaire. Details on measurement: The correlation will be evaluated using Pearson's correlation coefficient.

SECONDARY OUTCOMES:
The perceived benefits of psychological counseling throughout the care pathway. | 8 months
  This outcome will be assessed with an open question ("Do you think that the psychological sessions have helped support you along the care pathway? If yes, in which aspects of your experience was it helpful?"). Details on measurement: The perceived benefits of psychological counseling will be evaluated via open questions.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Pravettoni, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No